CLINICAL TRIAL: NCT01353365
Title: Surfactant Associated Protein - A Novel Marker for the Diagnosis of Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Gideon Berger, Rambam Health Care Campus
Other Study IDs: 0462-09/CTIL
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-04

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute dyspnea and chest discomfort are common complaints. Distinguishing between the entities that may present with such symptoms can be difficult. This project aims to study - venous thromboembolism (VTE) - a difficult diagnosis that can easily be missed yet its treatment is highly effective.

VTE represents a spectrum of disease ranging from deep vein thrombosis to pulmonary embolism (PE). Early diagnosis of PE is usually based on suspicion raised by clinical symptoms combined with a medical history of obvious predisposing factors. However, in around 30% of cases PE occurs in the absence of any predisposing factors. Individual clinical signs and symptoms are neither sensitive nor specific.

PE is generally associated with hypoxaemia, but up to 20% of patients with PE have a normal arterial oxygen pressure .Classic ECG changes are generally associated with the more severe forms of PE.

Bio-markers such as Plasma D-dimer (DD) have been investigated extensively in recent years. It has been shown that a normal DD level renders acute PE or DVT unlikely; on the other hand DD is not useful for confirming VTE.

CT angiography(CTA) has become the method of choice for imaging the pulmonary vasculature for suspected PE. Yet as in DD the pre-test probability of PE based on the clinician's abilities highly affects the results of the CT.

While VTE is a fairly common and sometimes lethal condition its diagnosis is difficult and based more on clinical hunches than on highly sensitive and specific diagnostic tools. It's quite evident that finding a novel, sensitive and even more importantly specific biomarker for PE would change the current approach and work-up needed for reaching a diagnosis.

We propose using serum levels of surfactant associated protein (SAP) as such a bio-marker. Surfactant is a unique phospholipoprotein secreted solely by type II alveolar cells in the lungs. About 90% of the surfactant structure is composed of phospholipids and the remaining 10% is composed of specific proteins.

Working hypothesis and aims: PE causes ischemic damage to lung tissue. Such damage will ultimately lead to a rise of serum SPA. The primary objective of this project is to ascertain the fact that indeed there is a rise of serum SPA among patients diagnosed with PE, what is the time-concentration profile of such rise and is the rise correlated to the size of the embolus.

Methods: The study will be designed as a prospective study consisting of several steps. The measurement of serum SPA will be done by commercially available ELISA kits. All patients will be enrolled by researchers from both the ER and internal B ward at the Rambam Medical Center.

Probable implications to Medicine: If indeed SPA levels will be proven to be a novel bio-marker for PE this could ultimately lead to a totally different approach in the classification and treatment of patients presenting with signs that may be associated with PE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven PE by CT- angiography or by V-Q scans (only high likelihood scans will be regarded as proven PE).

Exclusion Criteria:

* Under 18 years old.
* Unable to sign informed consent
* Other known pulmonary disease such as IPF, ARDS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with PE at ER and Internal B department at the Rambam Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-06

CONTACTS AND LOCATIONS:
Overall Officials: Berger Gideon, MD, Principal Investigator — Rambam Health Care Campus